CLINICAL TRIAL: NCT01627535
Title: Feasibility of Intraoperative Optical Imaging and Spectroscopy in Brain Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11320; NCI-2012-01074 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-06-20; First posted 2012-06-25 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Brain Tumor
Keywords: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Optical Imaging (Experimental): Patients undergo i2DOS
  Interventions: Other: Interoperative Optical Imaging and Spectroscopy

INTERVENTIONS:
Other: Interoperative Optical Imaging and Spectroscopy — Real time processing and display of i2DOS maps in the operating arena

SUMMARY:
This clinical trial studies optical imaging in assessing activity during surgery in patients with brain tumors. New procedures, such as optical spectroscopy, may help doctors maximally remove brain tumors and minimize damage to normal brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop the instrumentation to achieve real time processing and display of intraoperative 2-dimensional optical imaging and spectroscopy (i2DOS) maps in the operating arena.

II. To examine the timing and spatial involvement of human cortex intraoperatively to different stimuli using i2DOS.

OUTLINE: Patients undergo i2DOS.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical patient population in the City of Hope brain and spinal tumor neurosurgical programs that have been diagnosed with a brain tumor.
* Only lucid patients qualified to consent to neurosurgical procedure will be approached for participation in this study.
* We do intend to enroll subjects with potentially terminal brain tumors. Due to the potential benefit of intraoperative mapping, we are not planning to exclude these subjects.
* Patients with any type of brain tumor will be eligible for participation.
* All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* There are no exclusion criteria except for individuals without a brain tumor and the location of the craniotomy. If the exposed area of brain is not compatible with peripheral stimuli or volitional activity the subject cannot be enrolled.
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Determination of the effectiveness of intraoperative optical imaging technology and optical spectroscopy. | Day 1 post surgery
  Optical reflectance images will be analyzed by pixel by-pixel subtraction of a control trial and a stimulation trial. This subtracted image will then be divided by the control image to normalize for differences between subjects and trials. These ratios thus represent proportional changes from baseline.
Intraoperative determination of the location of critical brain functions. | Day 1 post surgery
  We will examine the timing and spatial involvement of human cortex intraoperatively to different stimuli using i2DOS. Stimulus parameters will be varied to investigate stimulus-response relationships. We will study areas of sensori-motor and language cortex using customary stimuli for evoked potentials (i.e. transcutaneous electrical nerve stimulation), tactile stimuli for exposed cortical dermatome representations, and language tasks for cortical language representations. Results will be correlated with intraoperative electrophysiological measures.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Prakash, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States